CLINICAL TRIAL: NCT07047313
Title: Impact of Adding Jones Technique to Mulligan Therapy in Patients With Cervicogenic Headache
Acronym: CGH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator : alshaymaa shaaban abd el azeim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005807
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cervicogenic Headache
Keywords: jones technique; mulligan therapy; cervicogenic headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: jones and mulligan therapy
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- jones and mulligan therapy (Experimental): thirty patients will receive the Jones technique puls mulligan and exercises programe three times a week for four weeks
  Interventions: Other: jones and mulligan therapy; Other: mulligan therapy; Other: exercises program
- mulligan therapy (Experimental): thirty patients will receive mulligan therapy and exercise programs three times a week for four weeks
  Interventions: Other: mulligan therapy; Other: exercises program
- exercises program (Active Comparator): thirty patients will receive exercise programs three times a week for four weeks
  Interventions: Other: exercises program

INTERVENTIONS:
Other: jones and mulligan therapy — for jones technique in upper trapezius and suboccipital muscles, the participants supine , the therapist used manual palpation to locate the tender area in the UT and sub-ossipital muscles. Once detected, pressure to the tender area was progressively increased . The participant was then repositioned passively to decrease the stress under palpation, resulting in a 70% subjective decrement in pain. That position was maintained for 90 s. eventually, the participant returned to the neutral position slowly and passively. for mulligan SNAGS,The therapist held the patient with his trunk, and wrapped the patient's head lightly with his arm on the patient's side, and placed the ring finger on the trouble spot right above the small vertebral joint. The therapist placed the thenar eminence of his opposite hand on the ring finger, which was touching the lesion site. On the site, the therapist performed gliding in the upward direction of the front pupil (45 degrees) exercises
  Arms: jones and mulligan therapy
Other: mulligan therapy — mulligan SNAGS,The therapist held the patient with his trunk, and wrapped the patient's head lightly with his arm on the patient's side, and placed the ring finger on the trouble spot right above the small vertebral joint. The therapist placed the thenar eminence of his opposite hand on the ring finger, which was touching the lesion site. On the site, the therapist performed gliding in the upward direction of the front pupil (45 degrees). The hand, which was touching the spinous process, should be relaxed in order not to squeeze too hard. The source of the power of gliding on the joint surface must come from the opposite hand of the patient-contacting hand. Gliding was applied rhythmically (three times per second) and the width of gliding starts from the middle to the end+ exercises
  Arms: jones and mulligan therapy; mulligan therapy
Other: exercises program — The exercise program will be in the form of stretching exercises for the sternocleidomastoids (SCM), the scalenes, and upper fibers of trapezius; strengthening isometric exercises for the neck flexors, extensors, lateral flexors, and neck rotators; and postural correction exercises.

SUMMARY:
this study will be conducted to investigate impact of adding jones technique to mulligan therapy in patients with cervicogenic headache

DETAILED DESCRIPTION:
Cervicogenic headache (CeH) is a secondary headache attributed to dysfunctions of the cervical spine (international headache society. CGH is a non-throbbing, unilateral, side locked headache that originates in the cervical spine and gradually spreads to the occipital, temporal and orbital areas. It is associated with neck pain or stiffness and is often aggravated by sustained neck postures, repeated neck movements or physical activity. A survey published in 2003 found that strain-counterstrain was the forth most commonly used manipulative technique among providers of osteopathy in the US. The most common explanation for the effects of strain-counterstrain is that it influences aberrant neuromuscular activity mediated by muscle spindles, local circulation and inflammatory reactions. Clinical research into the effects of strain-counterstrain has only begun to emerge in recent years . The Mulligan manoeuvre is one of the best manipulations. Unlike traditional mobilization, which relies solely on the therapist, Mulligan posited that by exerting pressure on the spinous processes in a weight-bearing stance, the facet joints would undergo a synchronized sliding motion in a parallel manner. At the same time, It requires the patient to move actively in order to achieve the perfect therapeutic effect ,The Mulligan maneuver is highly efective in the manipulative treatment of CEH A systematic review have demonstrated the efficacy of the Mulligan maneuvre for CEH on clinical pain scales and cervical range of motion after treatment

ELIGIBILITY:
Inclusion Criteria:

* 20 to 60 years old patient with unilaterally of the head pain
* pain triggered by external pressure over the upper cervical joints (c1-c3)
* pain elicited by the neck movements, and/or sustained awkward positions with reduced neck ROM
* headache intensity pain score of at least 20mm on the Visual analogue scale (VAS)
* headache frequency of at least once a week for at least 3 months
* minimum neck disability index score of 10 points or greater

Exclusion Criteria:

* Migraine, tension- type headache, tumor, osteoporosis, fracture, rheumatoid arthritis and metabolic diseases.
* Prolonged history of steroid use.
* Resting blood pressure greater than 140/90 mmhg.
* cervical spinal stenosis, diminished sensation and central nervous system involvement,
* previous head or neck surgery or whiplash injury history within the last 6 weeks

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
pain intesnity | up to four weeks
  visual analogue scale will be used to asses pain intensity which patient will be instructed to put point on line from no pain to tolerable pain. The scale consists of a line, usually 100 mm long, ranging from no pain or discomfort (zero) , to the worst pain that could possibly feel .
headache disability | up to four weeks
  The Headache spesific Disability Questionnaire was used to assess headcahe disability. it is a self-administered scale with 9 items that assesses pain intensity, work or school disruptions, and the effect on recreational activities in individuals with headache complaints. Higher scores reflect greater impairment.

SECONDARY OUTCOMES:
neck disability | up to four weeks
  will be measured by Arabic neck disability index. It contains ten category/classes. Each category contains six choices (zero-five).Score from zero to four no disability, from five to 15 this is mild, From 15 to 24 this is moderate, from 25 to 34 this is severe, more than 34 this is a complete disability
pressure pain threshold | up to four weeks
  pressure pain threshold pressure pain threshold will be assessed by commander algometer
cervical range of motion | up to four weeks
  range of motion will be measured by inclinometer CROM. The CROM (deluxe version - Performance Attainment Associates, Roseville, MN, USA) measures the cervical range of motion5- for fexion, extension, lateral fexion, and rotation using separate inclinometers. These inclinometers are attached to a frame similar to that for eyeglasses one in the sagittal plane for fexion - extension, second in the frontal plane for lateral fexion and a third in the horizontal plane for rotation.
headache frequency | up to four weeks
  the number of days the subjects feel headache (headache frequency).
medication intake | up to four weeks
  from the patients' diary in the last week , medications intake will be recorded as follow: 1) not at all; 2) once a week; 3) once every couple of days; 4) once or twice a day; or 5) three or more times a day
headache duration | up to four weeks
  the total hours of headache (headache duration).